CLINICAL TRIAL: NCT04174872
Title: A Comparative Study Between Dexmedetomidine and Midazolam as Adjuvant to Bupivacaine During Epidural Anesthesia For Elective Gynecological Operations
Brief Title: Epidural Anesthesia for Gynecological Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Abdelhaleem Abdelrahman, Lecturer of Anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ME-2001
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Epidural Analgesics for Comparison
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Other): It has a sedative effect without significant respiratory depression , anxiolytic, analgesic, antihypertensive and sympatholytic properties. It is now being used as a neuraxial adjuvant that can be used as an effective adjuvant in epidural anaesthesia as it intensifys the motor block and prolongs the duration of postoperative analgesia.
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam
- Midazolam (Other): Midazolam has been reported to have a spinally mediated analgesic effect. Clinically, single-shot epidural or spinal administration of midazolam has been shown to have an analgesic effect on perioperative pain.
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — it has a sedative effect without significant respiratory depression , anxiolytic, analgesic, antihypertensive and sympatholytic properties. It is now being used as a neuraxial adjuvant that can be used as an effective adjuvant in epidural anaesthesia as it intensifys the motor block and prolongs the duration of postoperative analgesia.
  Other Names: precedex
Drug: Midazolam — Midazolam has been reported to have a spinally mediated analgesic effect. Clinically, single-shot epidural or spinal administration of midazolam has been shown to have an analgesic effect on perioperative pain.

SUMMARY:
Regional anesthesia is the preferred mode of anesthesia for major abdominal surgeries in present times. Gynecological surgeries are often associated with severe pain requiring a well-planned analgesia regimen to ensure adequate patient-comfort, early mobilization, and to decrease stay time in the hospital/post-anesthesia care unit (PACU) enabling patients to return to their normal activities quicker. Dexmedetomidine has been approved by Food and Drug Administration (FDA) as a short-term sedative for mechanically ventilated intensive care unit (ICU) patients as it has a sedative effect without significant respiratory depression , anxiolytic, analgesic, antihypertensive and sympatholytic properties. Epidural administration of preservative free midazolam induces antinociceptive effects in humans, when midazolam is added it acts through gamma amino-butyric acid (GABA) receptors and enhances the affinity of GABA receptors. Midazolam is involved in the release of endogenous opioids acting on spinal delta receptors so antinociceptive effects of morphine like substances are potentiated when epidural midazolam is added. Studies have revealed that use of epidural midazolam provides effective analgesia in adults. So, the present study will evaluate the additive analgesic effects of epidural midazolam in combination with bupivacaine in elective gynecologic surgeries and compare the results with the use of bupivacaine with dexmedetomidine and observe the quality of epidural anesthesia with occurrence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of ASA I-II.
* Aged 18-55 years undergoing elective gynecological surgeries

Exclusion Criteria:

* Patient refusal.
* Patients with history of diabetes mellitus, cardiac disease, hypertension, chronic obstructive respiratory disease, coagulation abnormalities, spinal deformities, patients allergic to amide type of local anesthetics, localized skin sepsis, neurological disease, hepatic and renal diseases, peripheral neuropathy and psychiatric diseases.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Onset of sensory blockade | Eight months
  time interval from epidural injection of drugs to sensory blockade at T10

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Surgical ICU, and Pain Management, Cairo, Egypt